CLINICAL TRIAL: NCT03142282
Title: Maintenance Chemotherapy Versus Consolidative Radiotherapy Plus Maintenance Chemotherapy for Unresectable Metastatic Colorectal Cancer: A Randomized Phase II Trial
Brief Title: Consolidative Radiotherapy Plus Maintenance Chemotherapy for Metastatic Colorectal Cancer
Acronym: MCRC-LC1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Tao Zhang, Cancer Center, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCRC-LC1
Record Dates: First submitted 2017-04-26; First posted 2017-05-05 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Metastatic Colorectal Cancer; Radiotherapy
Keywords: maintenance treatment
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Maintenance Chemotherapy

STUDY DESIGN:
Intervention Model Description: Radiation: SBRT or IMRT Drug: Maintenance chemotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maintenance chemotherapy (Active Comparator): FDA approved drugs for the study population: Bevacizumab, Xeloda
  Interventions: Drug: maintenance chemotherapy
- Radiotherapy (Experimental): consolidative radiotherapy plus maintenance chemotherapy
  Interventions: Radiation: Consolidative Radiotherapy

INTERVENTIONS:
Drug: maintenance chemotherapy — National Comprehensive Cancer Network (NCCN) or European Society for Medical Oncology (ESMO) suggested maintenance chemotherapy regimens: xeloda, bevacizumab
  Arms: Maintenance chemotherapy
Radiation: Consolidative Radiotherapy — Stereotacticbodyradiationtherapy (SBRT) or intensity modulated radiation therapy (IMRT) for metastatic sites (less than 5)
  Arms: Radiotherapy

SUMMARY:
This study is a randomized phase II trial of maintenance chemotherapy versus consolidative radiotherapy plus maintenance chemotherapy for patients with unresectable metastatic colorectal cancer (MCRC).

DETAILED DESCRIPTION:
Prior to accrual on the trial, patients with unresectable metastatic colorectal cancer will be treated with palliative chemotherapy. And patients who achieve a partial response or stable disease by imaging criteria will receive maintenance chemotherapy. In our study, these group patients will be randomized to maintenance chemotherapy or consolidative radiotherapy to all sites of disease (followed by maintenance chemotherapy at the medical oncologist's discretion). Choices of palliative and maintenance chemotherapy will be determined by the medical oncologist based on clinical appropriateness.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have biopsy proven unresectable MCRC.
2. Patients must have received induction chemotherapy for 3-6 months, and achieved stable disease or a partial response.
3. Age ≥ 18 years
4. Patients must have measurable disease at baseline.
5. Patients can have up to only 5 discrete active extracranial lesions (≤3 in the liver and ≤3 in the lung) identified by position-emission tomography (PET) scan and also seen on correlative plain film, CT scan, or MRI within 8 weeks prior to the initiation of radiotherapy.
6. Patients who previously received radiotherapy to the primary site will be ineligible if there is CT evidence of disease progression within the past 3 months.
7. Patients must have a Karnofsky Performance Scores (KPS) >60
8. Aspartate aminotransferase, alanine aminotransferase & Alkaline phosphates must be ≤ 2.5 times the upper limit of normal (ULN). Total bilirubin must be within the limit of normal.
9. Patients should have adequate bone marrow function as defined by peripheral granulocyte count of ≥1500/mm³.
10. Patients should have adequate renal function (serum creatinine ≤1.5 times the ULN).
11. Females of childbearing potential should have a negative pregnancy test.
12. Patients who would be receiving radiation for lung lesions who are known or suspected by the treating radiation oncologist to have compromised lung function must have a documented forced expiratory volume in 1 second (FEV1) ≥ 1 litre.
13. Patients must provide verbal and written informed consent to participate in the study.
14. Total bilirubin: within normal institutional limits

Exclusion Criteria:

1. Patients with either untreated brain metastases or brain metastases treated within the past three months are ineligible
2. Patients with serious, uncontrolled, concurrent infection(s).
3. Significant weight loss (>10%) in the prior 3 months.
4. Treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cancers.
5. Patients with more than 5 discrete metastatic lesions.
6. Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
7. Unwillingness to participate or inability to comply with the protocol for the duration of the study.
8. Patients who are pregnant. Patients with reproductive capability will need to use adequate contraception during the time of participation in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2 years
  Evaluate the effect of consolidative radiotherapy with or without maintenance chemotherapy versus maintenance chemotherapy alone on progression free survival

SECONDARY OUTCOMES:
Actuarial rate in-field local control | 2 years
  To describe the actuarial rate in-field local control and rate of out-of-field disease progression
Toxicities | 2 years
  Acute toxicity was scored according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v3.0 criteria during and up to 3 months after radiotherapy. Late toxicity was graded using the Radiation Therapy Oncology Group (RTOG)/European Organisation for the Research and Treatment of Cancer (EORTC) criteria.
Overall survival | 5 years
  To evaluate overall survival after consolidative radiotherapy followed by maintenance chemotherapy in comparison to maintenance chemotherapy alone.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, MD,PHD, Study Chair — Cancer Center, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology , Wuhan 430022, China.
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Van Cutsem E, Cervantes A, Adam R, Sobrero A, Van Krieken JH, Aderka D, Aranda Aguilar E, Bardelli A, Benson A, Bodoky G, Ciardiello F, D'Hoore A, Diaz-Rubio E, Douillard JY, Ducreux M, Falcone A, Grothey A, Gruenberger T, Haustermans K, Heinemann V, Hoff P, Kohne CH, Labianca R, Laurent-Puig P, Ma B, Maughan T, Muro K, Normanno N, Osterlund P, Oyen WJ, Papamichael D, Pentheroudakis G, Pfeiffer P, Price TJ, Punt C, Ricke J, Roth A, Salazar R, Scheithauer W, Schmoll HJ, Tabernero J, Taieb J, Tejpar S, Wasan H, Yoshino T, Zaanan A, Arnold D. ESMO consensus guidelines for the management of patients with metastatic colorectal cancer. Ann Oncol. 2016 Aug;27(8):1386-422. doi: 10.1093/annonc/mdw235. Epub 2016 Jul 5. PMID 27380959
- [Result] Gomez DR, Blumenschein GR Jr, Lee JJ, Hernandez M, Ye R, Camidge DR, Doebele RC, Skoulidis F, Gaspar LE, Gibbons DL, Karam JA, Kavanagh BD, Tang C, Komaki R, Louie AV, Palma DA, Tsao AS, Sepesi B, William WN, Zhang J, Shi Q, Wang XS, Swisher SG, Heymach JV. Local consolidative therapy versus maintenance therapy or observation for patients with oligometastatic non-small-cell lung cancer without progression after first-line systemic therapy: a multicentre, randomised, controlled, phase 2 study. Lancet Oncol. 2016 Dec;17(12):1672-1682. doi: 10.1016/S1470-2045(16)30532-0. Epub 2016 Oct 24. PMID 27789196